CLINICAL TRIAL: NCT06179823
Title: Safety of Direct Oral Anticoagulant During Pregnancy - Pregnancy, Neonatal and Infant Outcome: a National-based Study From the French Claim Database
Brief Title: Safety of Direct Oral Anticoagulant During Pregnancy
Acronym: SACOD
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Aurélie BANNAY, MD, Central Hospital, Nancy, France
Other Study IDs: SACOD
Record Dates: First submitted 2023-12-12; First posted 2023-12-22 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Thromboembolic Disease
MeSH Terms: conditions — Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- DOAC direct oral anticoagulants: pregnant women exposed to doac
- VKA vitamin K antagonist: pregnant women exposed to vitamin K antagonist
- Heparin: pregnant women exposed to Heparin

SUMMARY:
Pregnancy is a major risk factor of thromboembolic disease (2 to 10 increased risk of thromboembolic event for pregnant women). This risk is related to the physiological changes inducing venous stasis and hypercoagulability.

Thromboembolic disease is the first preventable cause of death during pregnancy (in France 1.1 maternal death per 100 000 living births.

The recommended treatment for pregnant women is low molecular weight heparin requiring subcutaneous injections daily. Vitamin K antagonists are contraindicated due to a teratogenic risk. Direct oral anticoagulants (DOAC) are easier to use.

Currently available preclinical and incidental exposure data on DOAC in pregnant women are very limited and insufficient to conclude on their safety. Therefore, its use during pregnancy is currently contraindicated for the grounds of precaution. The use of reimbursement data from the Système National des données de santé (National Health Data System) would provide more information on accidental exposure to DOACs during pregnancy, thanks to its completeness.

The primary objective of SACOD is to compare the prevalence of adverse perinatal outcomes in pregnant women treated with a direct oral anticoagulant versus pregnant women treated with heparin and Vitamin K antagonist.

The secondary objectives of the SACOD study are to i) determine the frequency of patients exposed to a direct oral anticoagulant during pregnancy according to pregnancy, ii) measure the prevalence of adverse perinatal outcomes in pregnant women initiating treatment with a direct oral anticoagulant therapy, iii) compare the prevalence of adverse perinatal outcomes in pregnant women initiating treatment with direct oral anticoagulants compared with pregnant women treated with heparin and a vitamin K antagonist, iv) compare the prevalence of adverse perinatal outcomes in pregnant women with Antiphospholipid syndrome treated with a direct oral anticoagulant versus pregnant women treated with heparin and anti-vitamin K, v) measure the incidence of thrombo-embolic episodes during pregnancy under anticoagulant treatment.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women exposed to an anticoagulant

Exclusion Criteria:

* women not covered by national health insurrance

Ages: 10 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: All women with an pregnancy outcome identified in the French nationwide claim database (SNDS) exposed to anticoagulation treatment
Sampling Method: Probability Sample
Enrollment: 1755558 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Adverse pregnancy outcome | during pregnancy
  at least one of the following events :
  * miscarriage/aborption
  * termination of pregnancy,
  * stillbirth,
  * preterm birth,
  * death of a full-term newborn
Complication | from date of conception to the first year of child life
  at least one of the following events :
  * maternal complication (hemorrhage...)
  * child malformation

CONTACTS AND LOCATIONS:
Locations (1):
- Nancy teaching hospital, Nancy, France